CLINICAL TRIAL: NCT00918866
Title: A Phase IV, Open-Label Safety Evaluation of the Effect of DEFINITY® on Pulmonary Artery Hemodynamics in Patients With Normal and Increased Pulmonary Artery Pressure
Brief Title: A Study of Commercial DEFINITY® to Monitor the Effects of the Heart's Pulmonary Artery Pressure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lantheus Medical Imaging (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DMP 115-416
Record Dates: First submitted 2009-06-04; First posted 2009-06-11 (Estimated); Results first posted 2011-07-11 (Estimated); Last update posted 2020-11-24 (Actual); Status verified 2011-10

CONDITIONS: Pulmonary Heart Disease
Keywords: Phase 4; DEFINITY®; hemodynamics; pulmonary artery pressure
MeSH Terms: conditions — Pulmonary Heart Disease | interventions — perflutren

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low Pulmonary Arterial Pressure (Experimental): Subjects with pulmonary arterial pressure (PAP) of < or = to 35 mmHg.
  Interventions: Drug: Definity
- Elevated Pulmonary Arterial Pressure (Experimental): Subjects with a PAP of > or = to 35 mmHg.
  Interventions: Drug: Definity

INTERVENTIONS:
Drug: Definity — one bolus dose of Definity per intravenous injection, 30-60 second injection, dose value calculation = maximum of 10 microliter/kg patient weight
  Other Names: Perflutren Lipid Microsphere

SUMMARY:
The purpose of this clinical research is to learn if DEFINITY® 416 will cause any adverse effects during Right Heart Catheterization. This research was requested by the FDA.

DETAILED DESCRIPTION:
This Phase IV safety study will provide safety data on potential systemic and pulmonary hemodynamic effects caused by the administration of DEFINITY® in patients who are to undergo right heart cardiac catheterization for clinical reasons. Using a right heart catheter for direct measurements of pulmonary artery hemodynamics will allow accurate assessments of potential alterations of the pulmonary vasculature. This will be further investigated by the inclusion of two patient populations, one with a baseline pulmonary artery pressure < 35 mmHg, and one with elevated baseline pulmonary artery pressure. The addition of immune parameter measurements will assess a potential link between systemic and pulmonary alterations and potential immune reactions following DEFINITY® administration.

The inclusion of patients in this study is not based on a required echocardiogram with DEFINITY® administration because patients would be exposed to an unjustifiable risk of invasive right heart catheterization and are unlikely to consent to such a procedure. Therefore, patients undergoing heart catheterization for clinical reasons, or patients who are undergoing pulmonary artery hemodynamic assessments will be enrolled and receive DEFINITY® in this study.

ELIGIBILITY:
Inclusion Criteria:

* Appropriate candidate scheduled to undergo right heart catheterization and measurement of pulmonary artery hemodynamics for clinical reasons
* Be male or female above the age of 18
* Female patients who no longer have child-bearing potential
* Women of Child-Bearing Potential(WOCBP) who:

  1. are not pregnant and have been using an adequate and medically approved method of contraception
  2. have a negative urine pregnancy test
* Be able and willing to communicate effectively with study center personnel.

Exclusion Criteria:

* Women who are pregnant or lactating
* Known hypersensitivity or contraindication to or greater heart block
* Previous heart transplant
* Known right-to-left shunt (including atrial septal defect)
* Severe pulmonary artery hypertension (i.e., > 75 mmHg
* Current uncontrolled ventricular tachycardia
* Second-degree or greater heart block
* Any contraindications for the use of a right heart catheter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Lee, MD, Study Director — Lantheus Medical Imaging
Locations (8):
- United States (8):
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Methodist Hospital, Saint Louis Park, Minnesota
  - Cardiovascular Consultants, Kansas City, Missouri
  - Holy Name Hospital, Teaneck, New Jersey
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Health and Sciences University, Portland, Oregon
  - The University of Texas Medical Branch at Galveston, Galveston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: participants were recruited from hospitals and clinics in the USA between July 2009 and December 2009
Pre-assignment Details: There were no randomization procedures or other pre-assignment requirements in this study.
Period: Overall Study
Arm/Group | Low Pulmonary Arterial Pressure | Elevated Pulmonary Arterial Pressure
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Pulmonary Arterial Pressure | Elevated Pulmonary Arterial Pressure | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.9 (10.8) | 57.4 (15.1) | 57.2 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 17
  Male | 6 | 9 | 15
Pulmonary artery pressure 1 minute pre-dose [Mean (Standard Deviation); unit: mm Hg] | 30.4 (3.38) | 50.9 (10.31) | 40.7 (12.89)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Pulmonary Artery Pressure Change From 1 Minute Pre-dose to 31 - 35 Minutes Post Dose
Description: Percent change in pulmonary atery pressure change from immediately pre-dose to 31 - 35 minutes post dose
Time Frame: 31-35 minutes minus baseline
Population: Per the protocol
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Low Pulmonary Arterial Pressure | Elevated Pulmonary Arterial Pressure
Number analyzed (Participants) | 16 | 16
mm Hg | -1.9 (18.03) | -1.7 (10.25)

2. Secondary Outcome: Immunology Panel- Complement 3A (C3A)
Description: Evaluate the Immunology Panel after the administration of DEFINITY
Time Frame: Out to 70 minutes
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Low Pulmonary Arterial Pressure | Elevated Pulmonary Arterial Pressure
Number analyzed (Participants) | 15 | 15
ng/ml | -45.80 (338.14) | -38.20 (414.86)

3. Secondary Outcome: Immunology Panel- Complement 5A(C5A)
Description: Evaluate the Immunology Panel after the administration of DEFINITY
Time Frame: Out to 70 minutes
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Low Pulmonary Arterial Pressure | Elevated Pulmonary Arterial Pressure
Number analyzed (Participants) | 15 | 15
ng/ml | -0.95 (3.56) | 0.78 (4.55)

4. Secondary Outcome: Immunology Panel- Interleuken-6
Description: Evaluate the Immunology Panel after the administration of DEFINITY
Time Frame: Out to 70 minutes
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Low Pulmonary Arterial Pressure | Elevated Pulmonary Arterial Pressure
Number analyzed (Participants) | 14 | 11
pg/ml | 0.31 (1.46) | 0.15 (2.11)

5. Secondary Outcome: Immunology Panel- Tryptase
Description: Evaluate the Immunology Panel after the administration of DEFINITY
Time Frame: Out to 70 minutes
Measure: Mean (Standard Deviation); unit: ug/ml
Arm/Group | Low Pulmonary Arterial Pressure | Elevated Pulmonary Arterial Pressure
Number analyzed (Participants) | 16 | 14
ug/ml | -0.24 (0.82) | -0.01 (1.46)

ADVERSE EVENTS:
Time Frame: Through 32 hours
Arm/Group | Low Pulmonary Arterial Pressure | Elevated Pulmonary Arterial Pressure
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 4/16 | 5/16
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Pulmonary Arterial Pressure (N=16) | Elevated Pulmonary Arterial Pressure (N=16)
Chest Pain (General disorders) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No